CLINICAL TRIAL: NCT05493202
Title: Correlation of Urinary Estrone Glucuronide With Superovulatory Response in IVF Cycles.
Brief Title: Superovulation And Urinary Concentration of Estrone
Acronym: SAUCE
Status: Completed | Type: Observational
Sponsor: Olive Fertility Centre (Other)
Collaborators: Quanovate Tech Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SAUCE
Record Dates: First submitted 2022-08-02; First posted 2022-08-09 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: in Vitro Fertilization; Hormone Testing
Keywords: in vitro fertilization; IVF; hormone testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Study group: 30 patients undergoing gonadotropin stimulation for IVF or egg freezing.
  Interventions: Device: Mira Fertility Tracker

INTERVENTIONS:
Device: Mira Fertility Tracker — Non-interventional: observational, documenting urine E3G levels during gonadotropin stimulation.

SUMMARY:
To determine if measurement of urinary estrone glucuronide concentrations with an at-home device is correlated with superovulatory response during gonadotropin stimulated IVF cycles.

DETAILED DESCRIPTION:
Hypothesis

Urinary estradiol concentrations measured with an at-home device correlates with gonadotropin response during superovulation for IVF and can serve as an alternative to serum estradiol measurements.

Justification

The in vitro fertilization (IVF) process entails gonadotropin stimulation to obtain supernumerary oocytes. To ensure an adequate and safe administration, gonadotropin treatment requires monitoring with transvaginal sonography (TVS) to determine the quantity and size of ovarian follicles. In addition, serum estradiol (E2) concentration reflects bioactivity of the follicles and is used to modulate dosing. TVS and E2 are complementary modalities used synchronously to dynamically optimize the gonadotropin protocol. For the typical IVF stimulation cycle with an GnRH antagonist protocol, the patient will require 10-12 days of gonadotropin administration, during which time the 3-6 visits for TVS and blood tests will be needed.

Reducing the invasiveness of procedures can improve the patient experience. Repetitive phlebotomy, as is required for serum estradiol measurements during IVF, can be unpleasant and painful. Thus, a less invasive alternative with at-home urinary testing may be more desirable and convenient.

Estrone glucuronide (E3G) is a metabolite of E2 that can be measured in the urine. Urinary E3G with an FDA and CE registered home device called the Mira Fertility Tracker ("Mira"). Correlation between the serum hormones and their respective urinary metabolites has been established but the efficacy of monitoring urinary E3G has not been demonstrated in the context of IVF.

The purpose of the current observational study is to compare urinary E3G with traditional serum E2 monitoring during gonadotropin stimulation for IVF and correlate the levels with stimulation outcomes. If validated, urinary hormone monitoring could serve as a more patient-friendly alternative to repetitive phlebotomy required for serum hormone measurement during IVF.

Research Design

Patients will undergo IVF per clinical indication. Gonadotropin dosing will be determined at the discretion of the responsible physician using standard dosing criteria (age, ovarian reserve testing, prior history, etc). For consistency of comparison, the study population will focus on patients with a normal ovarian reserve (AMH 1-3.5ng/mL).

During stimulation, the monitoring schedule will be consistent with routine clinical protocols. In general, the initial E2 are determined on day 6 of stimulation from a single serum sample, and subsequent serum E2 and TVS are checked from day 8 onwards, as is clinically indicated by patient response to gonadotropin stimulation.

Urinary E3G will be monitored daily with first morning urine from the first day through the final day of gonadotropin stimulation. A Mira device and testing wands will be provided to each participating patient and urinary testing will be performed by the patient at home.

Primary outcomes will include correlation of E3G with the number of total and mature oocytes retrieved, and a comparison to the serum E2 correlation to the same parameters. Secondary outcomes will include correlation of urinary E3G and serum E2 levels throughout stimulation.

Additional details regarding laboratory study protocols are as follows:

Measurement of urine E3G: The Mira be used to measure urinary E3G via immunofluorescence method. First morning urine will be collected by the patient at home. A test wand will be dipped into the urine sample for ten seconds, then inserted into a palm-sized device.

All other protocols are consistent with routine clinical practice. Briefly, serum samples for E2 will be collected by venipuncture and processed using a commercially available E2 chemiluminescent assay on automated immunoanalyzer (Beckman-Coulter Access 2) in an accredited commercial laboratory (Novavita, Vancouver, BC). Sonography will be performed by licensed physicians with an endovaginal probe, consistent with standard clinical practice. IVF laboratory procedures will be performed by trained embryologists at the Olive Fertility Centre (Vancouver, BC).

ELIGIBILITY:
Inclusion Criteria:

Ages 21-45 AMH between 1-3.5 ng/mL (7.14-24.5 pmol/L) within 1 year of enrollment Gonadotropin stimulation with GnRH antagonist protocol Able to collect 1st morning urine

Exclusion Criteria:

Aversion to phlebotomy (as is normally required during IVF). Use of aromatase inhibitors during stimulation (which can affect serum E2 levels)

Ages: 21 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Females who are undergoing gonadotropin stimulation for IVF.
Study Population: Patients will be recruited from patients undergoing IVF or egg freezing at the Olive Fertility Centre.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-02-20 (Actual); Primary Completion 2022-06-13 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Correlation of E3G with oocyte retrieval parameters | Approximately 2 weeks per patient to complete data collection
  Regression of E3G levels to total and mature number of oocytes retrieved
Correlation of E3G and E2 levels throughout stimulation | Approximately 2 weeks per patient to complete data collection
  Comparison of urine and serum hormone levels

CONTACTS AND LOCATIONS:
Locations (1):
- Olive Fertility Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nakhuda GS, Li N, Yang Z, Kang S. At-home urine estrone-3-glucuronide quantification predicts oocyte retrieval outcomes comparably with serum estradiol. F S Rep. 2023 Jan 28;4(1):43-48. doi: 10.1016/j.xfre.2023.01.006. eCollection 2023 Mar. PMID 36959966